CLINICAL TRIAL: NCT01811966
Title: Preoperative Volume Substitution in Fasting Patients Undergoing Elective Surgery - Impact on Hemodynamic Stability During Anesthesia
Brief Title: Preoperative Volume Substitution in Elective Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Dr. Thomas Kratz, Dr. Thomas Kratz, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKGMVolume; UKGMVolume (Other: University Hospital of Marburg)
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Hemodynamic Instability; Hypovolemia; Anesthesia
Keywords: preoperative volume substitution; hypovolemia; preoperative fasting
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): preoperative none substitution of i.v. fluids.
  Interventions: Other: Control
- Volume (Active Comparator): preoperative substitution of a defined amount of i.v. fluids (8 ml/kg RingerAcetate solution for 15 min prior to introduction of anesthesia).
  Interventions: Other: Volume

INTERVENTIONS:
Other: Volume
  Other Names: RingerAcetate Solution; cristalloide
  Arms: Volume
Other: Control
  Arms: Control

SUMMARY:
Preoperative fasting can evoke a hypovolemia which may cause a hemodynamic instability during introduction of anesthesia.

The purpose of this study is to test the hypothesis that a defined preoperative volume substitution compared to standard procedure will result in a reduced incidence of hemodynamic instabilities during introduction of anesthesia in elective surgery patients.

DETAILED DESCRIPTION:
The preoperative fasting period often lasts longer than 2 hours as recommended by various national and international anesthetic guidelines. Thus, hypovolemia is more often then anticipated. In awake patients this condition is often masked. Introduction of anesthesia often leads to an unmasking of hypovolemia with a consecutive hemodynamic instability.

Aim of the study is to test the hypothesis that a preoperative volume substitution (8 ml/kg RingerAcetate Solution in 15 min. prior to introduction of anesthesia) reduces possible hemodynamic instabilities during initiation of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* thyreoid, parathyroid or gallbladder surgery
* general anesthesia

Exclusion Criteria:

* coronary artery disease
* congestive heart disease (≥ New York Heart Association (NYHA) 2)
* insulin dependent diabetes mellitus
* renal insufficiency (creatinine > 2,0 mg/dl)
* cerebrovascular disease
* severe hypertension (≥ antihypertensive drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
hemodynamic instability | at time of introduction of anesthesia
  Hemodynamic instability during induction of anesthesia (0-10 min), defined as at least one of the following:
  * Systolic blood pressure < 80 mmHg or decrease of 20% in preexistent hypertension
  * Mean blood pressure < 50 mmHg or decrease of 20% or > 20 mmHg in preexistent hypertension
  * Bradycardia < 45/min or decrease of 20% in preexistent bradycardia < 60/min.
  * Tachycardia > 120/min
  * Cardiac index < 2.0 l/min/m²

SECONDARY OUTCOMES:
Stroke volume index > 35 ml/m2 | at time of anesthesia
Stroke volume variation < 12 % | at time of anesthesia
Enddiastolic area (EDA) > 10 cm2 | at time of anesthesia
  transthoracic echocardiographic parasternal short axis enddiastolic area
inferior vana cava diameter (VCI) > 15 mm | at time of anesthesia
  transthoracic echocardiographic inferior vena cava diameter

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kratz, MD, Principal Investigator — Department of Anesthesia and Intensive Care Medicine, University Hospital Marburg, Germany
Locations (1):
- University Hospital of Marburg, Department of Anesthesia, Marburg, Germany